CLINICAL TRIAL: NCT05833477
Title: Tracing Changed Production of Red Blood Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-20064997
Record Dates: First submitted 2022-09-22; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Erythrocytosis; Erythropoiesis Abnormal
MeSH Terms: conditions — Polycythemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Recombinant human erythropoietin treatment three times per week for three weeks
  Interventions: Drug: Recombinant human erythropoietin

INTERVENTIONS:
Drug: Recombinant human erythropoietin — Recombinant human erythropoietin treatment three times per week for three weeks

SUMMARY:
In competitive sport, it is illegal to manipulate erythropoiesis. Manipulated erythropoiesis can indirectly be identified by atypical fluctuations in key haematological variables. However, this method also has limitations and as it is known that some athletes still manipulate erythropoiesis it is necessary to develop new and more sensitive detection methods.

The primary purpose of the study is to examine the importance of altered erythropoiesis for surface and intracellular erythrocyte proteins, the number of immature reticulocytes, and for the haematological characteristics of the erythrocyte, such as volume, haemoglobin concentration and concentration of glycosylated haemoglobin, to assess whether these can be used to identify changed erythropoiesis. Furthermore, the aim is to examine whether these parameters are affected by freezer storage of erythrocytes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* 18-40 years
* physical fitness rating more than 50ml/kg/min
* non-smokers
* blood pressure <130/90 mmHg
* hemoglobin concentration 7-10.5 mM.

Exclusion Criteria:

* Blood donor who has donated blood within the last three months
* Participation in other concurrent clinical trials
* To participate in competitive sport during or three months after the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Changes in CD71 expression | In the period from two weeks before treatment to three weeks after treatment
  Treatment induced changes in CD71 expression on red blood cells
Changes in CD35 expression | In the period from two weeks before treatment to three weeks after treatment
  Treatment induced changes in CD35 expression on red blood cells
Changes in CD47 expression | In the period from two weeks before treatment to three weeks after treatment
  Treatment induced changes in CD47 expression on red blood cells
Changes in CD55 expression | In the period from two weeks before treatment to three weeks after treatment
  Treatment induced changes in CD55 expression on red blood cells
Changes in CD59 expression | In the period from two weeks before treatment to three weeks after treatment
  Treatment induced changes in CD59 expression on red blood cells
Changes in RNA expression | In the period from two weeks before treatment to three weeks after treatment
  Treatment induced changes in RNA expression in red blood cells
Changes in Mean Cell Volume | In the period from two weeks before treatment to three weeks after treatment
  Treatment induced changes in Mean Cell Volume distribution of red blood cells

SECONDARY OUTCOMES:
Changes in HbA1c | In the period from two weeks before treatment to three weeks after treatment
  Treatment induced changes in HbA1c content of red blood cells
Continous blood glucose levels | In the period from two weeks before treatment to three weeks after treatment
  Continuous blood glucose level throughout the study
Changes in CD71 cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  CD71 expression on red blood cells before and after cryopreservation
Changes in CD35 cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  CD35 expression on red blood cells before and after cryopreservation
Changes in CD47 cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  CD47 expression on red blood cells before and after cryopreservation
Changes in CD55 cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  CD55 expression on red blood cells before and after cryopreservation
Changes in CD59 cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  CD59 expression on red blood cells before and after cryopreservation
Changes in RNA cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  RNA expression inred blood cells before and after cryopreservation
Changes in Mean Cell Volume cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  Mean Cell Volume distribution of red blood cells before and after cryopreservation
Changes in Ferritin | In the period from two weeks before treatment to three weeks after treatment
  Quantification of plasma ferritin concentration
Changes in Complete Blood Count on Advia | In the period from two weeks before treatment to three weeks after treatment
  Complete Blood Count analysis on the Advia 2120i instrument
Changes in Complete Blood Count on Sysmex | In the period from two weeks before treatment to three weeks after treatment
  Complete Blood Count analysis on the Sysmex XN-450 instrument
Changes in Complete Blood Count on Advia - cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  Complete Blood Count analysis on the Advia 2120i instrument before and after cryopreservation
Changes in Complete Blood Count on Sysmex - cryopreserved | Cryopreserved cells are measured 6 months after sample collection
  Complete Blood Count analysis on the Sysmex XN-450 instrument before and after cryopreservation
Changes in ALAS 2 | Up to 5 years
  Quantification of ALAS 2 in dried blood spots stored at room temperature, -20C and -80C
Changes in CA1 | Up to 5 years
  Quantification of CA1 in dried blood spots
Changes in SLC4a1 | Up to 5 years
  Quantification of SLC4a1 in dried blood spots
Changes in CD71 in dried blood spots | Up to 5 years
  Quantification of CD71 in dried blood spots
Changes in FECH | Up to 5 years
  Quantification of FECH in dried blood spots
Changes in Band 3 | Up to 5 years
  Quantification of Band 3 in dried blood spots
Changes in blood volume | Within 14 days before treatment and within 14 days after treatment
  Measurement of blood volume by CO rebreathing

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bejder, Ph.D., Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No